CLINICAL TRIAL: NCT01776723
Title: A Sequential Two-Stage Dose Escalation Study to Evaluate the Safety and Efficacy of Ruxolitinib for the Treatment of Chronic Myelomonocytic Leukemia (CMML) and Cataloging the Molecular Consequences of JAK2 Inhibition in Chronic Myelomonocytic Leukemia: A Correlative Study Identifying Targetable CMML Sub-Clones by Leveraging GM-CSF Dependent pSTAT Hypersensitivity
Brief Title: A Sequential Two-Stage Dose Escalation Study to Evaluate the Safety and Efficacy of Ruxolitinib
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-17259
Record Dates: First submitted 2013-01-24; First posted 2013-01-28 (Estimated); Results first posted 2020-03-12 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Myelomonocytic Leukemia
Keywords: Chronic Myelomonocytic Leukemia; CMML; Leukemia
MeSH Terms: conditions — Leukemia, Myelomonocytic, Chronic; Leukemia | interventions — ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- I: Dose Escalation - Ruxolitinib (Experimental): Phase I: Dose Escalation. In Phase I, participants will be allocated to dose levels starting at 10 mg/d (twice a day [BID] dosing) according to the "rolling six" Phase I design.
  Interventions: Drug: Ruxolitinib
- II: Maximum Tolerated Dose - Ruxolitinib (Experimental): Phase II: Treatment at Maximum Tolerated Dose (MTD).
  Interventions: Drug: Ruxolitinib

INTERVENTIONS:
Drug: Ruxolitinib — In Phase I, participants will be allocated to twice a day (BID) doses of 10 mg/d up to 40mg/d. The starting dose will be 10 mg/d (5mg BID). Each cohort will include up to 6 subjects. Once MTD is reached, 10 additional participants will be treated during the first stage of Phase II (stage 1) at the MTD.
  Other Names: Jakafi®; INCB-018424; Kinase Inhibitor

SUMMARY:
The purpose of this study is to find out if treating Chronic Myelomonocytic Leukemia (CMML) with a study drug [ruxolitinib] can improve outcomes of patients with CMML. The first step of the study is to learn the dose of ruxolitinib that is tolerable (bearable). It has already been studied in a number of patients with different bone marrow diseases and is approved for the treatment of a disease called Myelofibrosis; however, it is not approved for treatment of CMML. It is given orally (by mouth). Most people tolerate it well but the tolerability has not been determined in patients with CMML. We will be testing different doses to determine how much of the medication people can tolerate (bear) before they develop side effects.

DETAILED DESCRIPTION:
This is a phase 1/2, two-stage, sequential cohort dose escalation study. If dose escalation is completed as planned, no more than 53 subjects are expected to enroll onto this study at a rate of approximately 3 subjects every month. For the Phase 2 study the Simon's optimal two-stage design will be employed to test the null hypothesis that response rate (RR) equals to 10% versus the alternative that RR equals to 30%.

Demographic and clinical variables for the study patients will be summarized using descriptive statistics (mean, standard deviation, median, inter-quartile range, range, and frequency counts and percentages). Safety and efficacy data will be analyzed overall as well as separately for each dose cohort when appropriate.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of CMML using the World Health Organization (WHO) classification
* Age >18 years at the time of obtaining informed consent
* Must be able to adhere to the study visit schedule and other protocol requirements
* Must be able to provide adequate bone marrow (BM) aspirate and biopsy specimens for histopathological analysis and standard cytogenetic analysis during the screening procedure
* An Eastern Cooperative Oncology Group (ECOG) performance status score of 0,1, or 2
* Women of childbearing potential must have a negative pregnancy test at time of screening and baseline visits and agree to use two reliable forms of contraception simultaneously or to practice complete abstinence from heterosexual intercourse 1) for at least 28 days before starting study drug; 2) while participating in the study; and 3) for at least 28 days after discontinuation from the study.
* Must understand and voluntarily sign an informed consent form
* Must have a life expectancy of greater than 3 months at time of screening

Exclusion Criteria:

* Platelet count of less than 35,000/uL
* Absolute Neutrophil Count (ANC) of less than 250/uL
* Serum Creatinine >2.0
* Serum total bilirubin >1.5 x upper limit of normal (ULN)
* Use of cytotoxic chemotherapeutic agents, or experimental agents (agents that are not commercially available) for the treatment of CMML within 28 days of the first day of study drug treatment
* Any serious medical condition or psychiatric illness that will prevent the subject from signing the informed consent form or will place the subject at unacceptable risk if he/she participates in the study
* Concurrent use of Granulocyte/macrophage colony stimulating factor (GM-CSF). Granulocyte colony-stimulating factor (G-CSF) could be used for the short-term management of neutropenic infection. Stable doses of erythropoietin stimulating agents that were started >8 weeks from first ruxolitinib dose or corticosteroids that were being administered prior to screening are allowed.
* Uncontrolled current illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because ruxolitinib has not been studied in pregnant subjects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with ruxolitinib, breastfeeding should be discontinued if the mother is treated with ruxolitinib.
* Patients who have participated in other interventional (treatment-related) clinical trials within 30 days of enrollment are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-02-20 (Actual); Primary Completion 2018-11-28 (Actual); Study Completion 2022-05-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Padron, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (6):
- United States (6):
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Johns Hopkins Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Weill Medical College of Cornell, New York, New York
  - Cleveland Clinic, Cleveland, Ohio

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1, Level 1: Ruxolitinib 10 mg: Phase 1, Level 1: Ruxolitinib 5 mg twice daily
- Phase 1 Level 2: Ruxolitinib 20 mg: Phase 1 Level 2: Ruxolitinib 10 mg twice daily
- Phase 1 Level 3: Ruxolitinib 30 mg: Phase 1 Level 3: Ruxolitinib 15 mg twice daily
- Phase 1 Level 4: 40 mg Ruxolitinib: Phase 1 Level 4: 20 mg Ruxolitinib twice daily
- Phase 2: Maximum Tolerated Dose - Ruxolitinib: Phase II: Treatment at Maximum Tolerated Dose (MTD).
Period: Overall Study
Arm/Group | Phase 1, Level 1: Ruxolitinib 10 mg | Phase 1 Level 2: Ruxolitinib 20 mg | Phase 1 Level 3: Ruxolitinib 30 mg | Phase 1 Level 4: 40 mg Ruxolitinib | Phase 2: Maximum Tolerated Dose - Ruxolitinib
Started | 6 | 4 | 5 | 5 | 30
Completed | 6 | 4 | 5 | 5 | 30
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Phase 1, Level 1: Ruxolitinib 10 mg: Phase 1 Level 1: Ruxolitinib 5 mg twice daily
- Phase 1, Level 2: Ruxolitinib 20 mg: Phase 1 Level 2: Ruxolitinib 10 mg twice daily
- Phase 1, Level 3: Ruxolitinib 30 mg: Phase 1 Level 3: Ruxolitinib 15 mg twice daily
- Phase 1, Level 4: Ruxolitinib 40 mg: Phase 1 Level 4: Ruxolitinib 20 mg twice daily
- Phase 2: Maximum Tolerated Dose - Ruxolitinib: Phase 2: Treatment at Maximum Tolerated Dose (MTD).
- Total: Total of all reporting groups
Arm/Group | Phase 1, Level 1: Ruxolitinib 10 mg | Phase 1, Level 2: Ruxolitinib 20 mg | Phase 1, Level 3: Ruxolitinib 30 mg | Phase 1, Level 4: Ruxolitinib 40 mg | Phase 2: Maximum Tolerated Dose - Ruxolitinib | Total
Number analyzed (Participants) | 6 | 4 | 5 | 5 | 30 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 3 | 0 | 8 | 14
  >=65 years | 4 | 3 | 2 | 5 | 22 | 36
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 2 | 0 | 14 | 19
  Male | 5 | 2 | 3 | 5 | 16 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 4 | 5
  Not Hispanic or Latino | 6 | 4 | 4 | 4 | 26 | 44
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 6 | 4 | 5 | 5 | 29 | 49
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 6 | 4 | 5 | 5 | 30 | 50

OUTCOME MEASURES:

1. Primary Outcome: The Maximum Tolerated Dose (MTD) of Ruxolitinib for the Treatment of Myelomonocytic Leukemia (CMML)
Description: Phase I - The MTD is defined as the highest dose where less than 33% of participants experience a drug related predefined dose limited toxicity (DLT). Dose-limiting toxicity (DLT) is defined as any grade 4 hematologic toxicity and any grade 3 or greater non-hematologic toxicity except nausea that is controlled by antiemetic therapy based on the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. Grade 3 metabolic/electrolyte abnormalities that are not clinically significant, and are adequately controlled within 72 hours are not to be considered a DLT.
Time Frame: 17 weeks
Measure: Number; unit: mg
Arm/Group | I: Dose Escalation - Ruxolitinib
Number analyzed (Participants) | 20
mg | 40

2. Primary Outcome: Occurrence of Clinical Response
Description: Phase II - Proportion of participants achieving clinical benefit defined as hematologic improvement, complete remission (CR), partial remission (PR), marrow complete remission (Marrow CR) or stable disease (SD) by the International Working Group (IWG) 2006 criteria. Erythroid Response for pretreatment hemoglobin < 11 g/dl; Platelet response for subjects with a pre-treatment platelet count < 50 x 10^9/L; Neutrophil response with pretreatment absolute neutrophil count (ANC) < 1 x 10^9/L.
Time Frame: Up to 2 years
Population: All participants who received ruxolitinib therapy
Measure: Number; unit: participants
Arm/Group | II: Maximum Tolerated Dose - Ruxolitinib
Number analyzed (Participants) | 30
participants | 18

3. Secondary Outcome: Percentage of Participants With Acute Myeloid Leukemia (AML) Transformation
Description: Phase II - To determine the time to AML transformation of participants on Ruxolitinib. Acute myeloid leukemia (AML) transformation according to World Health Organization (WHO) criteria. CMML-1: peripheral blood <5% blasts, bone marrow <10% myeloblast. CMML-2: peripheral blood <19 percent blasts persistent monocytosis >1000/ul +/- cytopenias Leukocytosis frequent, bone marrow <19 percent blasts >10% dysplasia in affected lineage, Auer Rods.
Time Frame: Up to 2 years
Measure: Number; unit: percentage of patients
Groups:
- All Participants: All participants who received at least one dose of Ruxuxolitinib
Arm/Group | All Participants
Number analyzed (Participants) | 30
percentage of patients | 14

4. Secondary Outcome: Median Overall Survival (OS)
Description: Phase II - To determine the median overall survival.
Time Frame: Up to 2 years
Population: All participants who received ruxolitinib therapy
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | II: Maximum Tolerated Dose - Ruxolitinib
Number analyzed (Participants) | 30
months | 23.7 [13.3 to 30]

5. Secondary Outcome: Duration of Response in Days
Description: Phase II - To determine the duration of response achieved as in secondary endpoint one. The duration of response is measured from the time measurement criteria are met for major or complete platelet response (which ever is first recorded) until the first date that disease progression defined by the bone marrow response outlined above, progression/relapse following a CR, marrow CR or PR, or progressions/relapse following hematological improvement (HI) as outlined above.
Time Frame: 3.5 years
Measure: Mean (Full Range); unit: days
Groups:
- Phase 1, Level 2: Ruxolitinib 20 mg: Phase 1, Level 2: Ruxolitinib 10 mg twice daily
- Phase 1, Level 4: Ruxolitinib 40 mg: Phase 1, Level 4: Ruxolitinib 20 mg twice daily
- Maximum Tolerated Dose - Ruxolitinib: Treatment at Maximum Tolerated Dose (MTD).
Arm/Group | Phase 1, Level 1: Ruxolitinib 10 mg | Phase 1, Level 2: Ruxolitinib 20 mg | Phase 1, Level 3: Ruxolitinib 30 mg | Phase 1, Level 4: Ruxolitinib 40 mg | Maximum Tolerated Dose - Ruxolitinib
Number analyzed (Participants) | 6 | 4 | 5 | 5 | 30
days | 104 [55 to 172] | 446.25 [28 to 961] | 718 [54 to 1248] | 331.25 [60 to 853] | 263.5 [6 to 874]

ADVERSE EVENTS:
Time Frame: Adverse Events collected from time of consent through follow-up, up to 2 years
Groups:
- Phase 1, Level 2: Ruxolitinib 20 mg: Phase 1, Level 1: Ruxolitinib 10 mg twice daily
- Phase 1, Level 3: Ruxolitinib 30 mg: Phase 1, Level 1: Ruxolitinib 15 mg twice daily
- Phase 1, Level 4: Ruxolitinib 40 mg: Phase 1, Level 1: Ruxolitinib 20 mg twice daily
Arm/Group | Phase 1, Level 1: Ruxolitinib 10 mg | Phase 1, Level 2: Ruxolitinib 20 mg | Phase 1, Level 3: Ruxolitinib 30 mg | Phase 1, Level 4: Ruxolitinib 40 mg | II: Maximum Tolerated Dose - Ruxolitinib
All-Cause Mortality (participants affected / at risk) | 6/6 | 4/4 | 1/5 | 1/5 | 13/30
Serious Adverse Events (participants affected / at risk) | 6/6 | 4/4 | 1/5 | 1/5 | 15/30
Other Adverse Events (participants affected / at risk) | 6/6 | 4/4 | 5/5 | 5/5 | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1, Level 1: Ruxolitinib 10 mg (N=6) | Phase 1, Level 2: Ruxolitinib 20 mg (N=4) | Phase 1, Level 3: Ruxolitinib 30 mg (N=5) | Phase 1, Level 4: Ruxolitinib 40 mg (N=5) | II: Maximum Tolerated Dose - Ruxolitinib (N=30)
Facial muscle weakness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Death NOS (General disorders) | 6 (6) | 4 (4) | 1 (1) | 1 (1) | 13 (13)
Nervous system disorders - other (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Intracranial mass
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spleen disorder (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vascular disorders -Other (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Heart failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Respiratory, thoracic and mediastinal disorders - other (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infections and infestations - other (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Cellulitis on knee
Headache (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Multi-organ failure (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Surgical and medical procedures -other (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — knee replacement
Edema limbs (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal disorders - other (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — peptic ulcer bleeding
Surgical and medical procedures - other (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Orthopedic surgery on left humerus
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flu like symptoms (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1, Level 1: Ruxolitinib 10 mg (N=6) | Phase 1, Level 2: Ruxolitinib 20 mg (N=4) | Phase 1, Level 3: Ruxolitinib 30 mg (N=5) | Phase 1, Level 4: Ruxolitinib 40 mg (N=5) | II: Maximum Tolerated Dose - Ruxolitinib (N=30)
Fatigue (General disorders) | 3 (3) | 3 (5) | 4 (4) | 1 (1) | 10 (11)
Edema limbs (General disorders) | 3 (4) | 3 (4) | 1 (1) | 1 (1) | 4 (4)
Fever (General disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (2) | 8 (8)
Pain (General disorders) | 1 (1) | 1 (2) | 2 (4) | 0 (0) | 4 (6)
Chills (General disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (2) | 2 (2)
Non-cardiac chest pain (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 4 (5)
Flu-like symptoms (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Edema trunk (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Irritability (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Multi-organ failure (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 3 (11) | 2 (5) | 2 (3) | 5 (5)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 6 (6)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 6 (8)
Vomitting (Gastrointestinal disorders) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 3 (3)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 4 (5)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 5 (6)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Bloating (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Gastroparesis (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (2)
Hemorrhoids (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Esophageal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fecal incontinence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Malabsorption (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rectal hemorrhate (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (6) | 2 (2) | 1 (1) | 8 (11)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (8) | 2 (5) | 0 (0) | 9 (11)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 4 (6)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (5) | 1 (2) | 1 (2) | 4 (4)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchial stricture (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 2 (4) | 3 (4) | 2 (2) | 17 (24)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 2 (3) | 0 (0) | 9 (9)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 9 (15)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 2 (3) | 0 (0) | 7 (9)
Syncope (Nervous system disorders) | 1 (2) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (5)
Parathesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Movements involuntary (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Brachial plexopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Concentration impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Dysesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Facial muscle weakness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Meningismus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spasticity (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (2) | 2 (3) | 2 (2) | 1 (1) | 11 (17)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (3) | 3 (6) | 0 (0) | 7 (11)
Creatinine increased (Investigations) | 0 (0) | 2 (4) | 2 (3) | 0 (0) | 5 (8)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (2) | 3 (4) | 0 (0) | 3 (5)
Alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 4 (4)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (5)
Weight gain (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
White blood cell decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 1 (1)
Cardiac troponin I increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 3 (5) | 0 (0) | 6 (9)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 3 (4)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 2 (5) | 2 (3) | 0 (0) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 5 (11)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Acideosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 0 (0) | 2 (7) | 2 (6) | 1 (1) | 7 (12)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 6 (10)
Bronchial infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Skin Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 2 (3)
Bladder infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Papulopustular rash (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pleural infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Vaginal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Abdominal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mucosal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ottis media (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2) | 1 (3) | 2 (2) | 5 (9)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 7 (8)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 5 (5)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 3 (4)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Erythroderma (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypohidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 7 (7)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (2) | 2 (3) | 0 (0) | 6 (7)
Insomnia (Psychiatric disorders) | 3 (3) | 1 (1) | 1 (2) | 0 (0) | 5 (6)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hot flashes (Vascular disorders) | 0 (0) | 1 (1) | 1 | 0 (0) | 2 (2)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
Hematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphedema (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial fibillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Sinus tachycardia (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Heart failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 | 0 (0) | 0 (0) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Urinary urgency (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Urine discoloration (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Renal calculi (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blurred vision (Eye disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Watering eyes (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Middle ear inflammation (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Testicular disorder (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neoplasms benign, malignant or unspecified -Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Immune system disorders -Other (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Surgical and medical procedures - Other (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3)
Ear and labyrinth disorders -Other (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Eye disorders -Other (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Renal and urinary disorders -Other (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cardiac disorders - Other (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 | 3 (4)
Vascular disorders - Other (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Psychiatric disorders -Other (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Injury, poisoning and procedures complications - Other (Injury, poisoning and procedural complications) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders -other (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 1 (5) | 0 (0) | 6 (7)
Musculoskeletal and connective tissue disorder -Other (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Infections and infestations - Other (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 6 (9)
Metabolism and nutrition disorders -Other (Metabolism and nutrition disorders) | 1 (1) | 3 (7) | 2 (4) | 0 (0) | 1 (1)
Investigations - Other (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Nervous system disorders -Other (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Blood and lymphatic system disorders - other (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 4 (4)
Respiratory, thoracic and mediastinal disorders - other (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 5 (5)
Gastrointestinal disorders - other (Gastrointestinal disorders) | 1 (2) | 1 (2) | 2 (3) | 0 (0) | 4 (6)
General disorders and administration site conditions - other (General disorders) | 1 (1) | 0 (0) | 3 (4) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-28): https://cdn.clinicaltrials.gov/large-docs/23/NCT01776723/Prot_SAP_000.pdf